CLINICAL TRIAL: NCT06317818
Title: Is Local Injection of Mesenchymal Stem Cells After Endoscopic Dilation Safe and Does it Improve the Outcome of Intestinal Stricture in Patients With Crohn's Disease?
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Sophie Vieujean, Head of Clinic, Centre Hospitalier Universitaire de Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJT2301
Record Dates: First submitted 2024-02-08; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Safety Issues; Efficacy

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "MSCs" group (Experimental): One local injection of MSCs (3*10^7 cells) after endoscopic dilatation of the stricture
  Interventions: Other: Mesenchymal Stem Cells
- "control" group (Placebo Comparator): One local injection of the placebo (cell-free cell suspension solution devoid of cells) after endoscopic dilatation of the stricture
  Interventions: Other: Comparative placebo

INTERVENTIONS:
Other: Mesenchymal Stem Cells — Suspension of mesenchymal stromal cells for intratissular injection
  Arms: "MSCs" group
Other: Comparative placebo — Cell-free cell suspension solution devoid of cells for intratissular injection
  Arms: "control" group

SUMMARY:
This is an exploratory phase II study, to evaluate the impact of these Mesenchymal Stem Cells (MSCs) on strictures in Crohn's disease patients with symptomatic intestinal stricture eligible to endoscopic dilatation. The impact of combined treatment by endoscopic dilation and local injection of MSCs will be compared with that of a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years with Crohn's Disease diagnosed more than 6 months ago
* Background treatment, for Crohn's Disease, stable for 4 months
* Presence of stricture (whether de novo or anastomotic), meeting the radiological definition of stenosis, i.e. a combination of the following criteria: (1) localized luminal narrowing (reduction of luminal diameter by at least less than 50% compared to adjacent healthy bowel segment), (2) bowel wall thickening (25% increase in wall thickness compared to adjacent unaffected bowel) and pre-stenotic dilation (luminal diameter greater than 3 cm)
* Presence of symptomatic stricture with abdominal pain after meals and limitations on the amount or type of food at screening
* Presence of a stenosis accessible by ileo-colonoscopy, not passable (i.e. not allowing the passage of the adult ileo-colonoscope), of a length less than 5 cm, eligible for endoscopic dilation
* Patient accepting the study protocol and having signed an informed consent
* Patient capable of undergoing entero-MRI

Exclusion Criteria:

* Patient liable for immediate surgery
* Patient with intra-abdominal fistula or abscess
* Patient with a stenosis not accessible to ileocolonoscopy
* Patient presenting ≥ 2 strictures with impossibility of determining which stenosis is "dominant" and responsible for the symptoms (based on dilation in entero-MRI)
* Patient with a stenosis longer than 5 cm
* Patient with a contraindication to performing an entero-MRI or to the use of contrast product injection in entero-MRI (Gadolinium)
* Pregnant woman or planning a pregnancy in the year
* Patient with kidney insufficiency (with anuria, glomerular filtration rate < 30 ml/min or on dialysis), hepatic insufficiency (presence of fulminant hepatitis, cirrhosis with signs of portal hypertension, acute alcoholic hepatitis, esophageal varices, history of gastrointestinal bleeding following rupture of esophageal varices, hepatic encephalopathy, prolonged prothrombin time, ascites secondary to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with a total serum bilirubin level > 3 mg/dL)
* Patient with documented human immunodeficiency virus (HIV) infection, active hepatitis B or C or tuberculosis
* Patient having presented an opportunistic infection in the 6 months preceding inclusion or a serious infection in the previous 3 months
* Patient who has developed a malignant tumor with a history of lymphoproliferative disease with the exception of: non-melanoma skin cancer, carcinoma in situ (e.g. skin, cervix, bladder, breast) and in remission for at least 3 years prior to screening, superficial bladder cancer, asymptomatic low-grade or localized curatively treated prostate cancer for which the "watch-and-wait" approach is the standard of care as well as any other cancer that has been in remission for ≥ 3 years prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety of local MSCs injection, in association with endoscopic dilation, in strictures of patients with Crohn's disease. | From Week 0 to Week 48
  Recording of occurrence of adverse events (serious or not) up to week 48
Assessment of efficacy of local MSCs injection, in association with endoscopic dilation, in strictures of patients with Crohn's disease by evaluating symptomatic clinical response | Between Week 0, Week 24 and Week 48
  The symptomatic clinical response will be assessed by a composite score, calculated over an average of 7 days, taking up 2 of the 16 questions of the S-PRO or Stenosis Patient Reported Outcome in English (also called Stricturing Crohn's Disease Questionnaire). A score for postprandial abdominal pain < 2 and an average score, out of 7 days, for amount of types of food <2 also.
Assessment of efficacy of local MSCs injection, in association with endoscopic dilation, in strictures of patients with Crohn's disease by evaluating endoscopic response | Between Week 0, Week 24 and Week 48
  The endoscopic response will be defined by the ability to pass an adult colonoscope (complete endoscopic response) or an increase in lumen diameter (partial endoscopic response) measured in comparison with the size of an open biopsy forceps (7mm)
Assessment of efficacy of local MSCs injection, in association with endoscopic dilation, in strictures of patients with Crohn's disease by evaluating radiological response | Between Week 0, Week 24 and Week 48
  The radiological response will be defined by the presence of 3 of the 4 following criteria: (1) an improvement in luminal narrowing (improvement greater than 50% and/or reduction in luminal diameter of less than 50%); (2) improvement in pre-stenotic dilation (pre-stenotic dilation reduced by 50%, bowel diameter equal to normal bowel and/or pre-stenotic dilation improved to less than 2.5 cm); (3) reduction in wall thickening (50% improvement in gut wall thickening); (4) a reduction in the length of the stricture (50% improvement)

SECONDARY OUTCOMES:
Evaluation of studying, in addition to biomarkers (CRP and fecal calprotectin), | Weeks 0, 4, 12, 24, 36 and 48
  Evaluation of evolution of biomarkers (CRP and fecal calprotectin) over the time by blood and stool samples analysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium